CLINICAL TRIAL: NCT00108368
Title: The Cognitive Effects of Risperidone and Olanzapine
Brief Title: The Effects of Risperidone and Olanzapine on Thinking
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: US Department of Veterans Affairs (U.S. Federal Agency)
Collaborators: Janssen, LP (Industry)
Organization: VA Office of Research and Development (U.S. Federal Agency)
Allocation: Randomized | Model: Single Group | Masking: Double | Purpose: Treatment
Other Study IDs: MHBS-057-00S
Record Dates: First submitted 2005-04-14; First posted 2005-04-15 (Estimated); Last update posted 2009-01-21 (Estimated); Status verified 2007-09

CONDITIONS: Schizophrenia; Psychotic Disorders
Keywords: schizophrenia; cognition; antipsychotic medication; information processing; social cognition; Psychotic
MeSH Terms: conditions — Schizophrenia; Psychotic Disorders; Mental Disorders | interventions — Risperidone; Olanzapine

INTERVENTIONS:
Drug: Risperidone
Drug: Olanzapine

SUMMARY:
The goal of this research is to find ways to maximize the benefits of antipsychotic medications for cognition.

Hypothesis: Risperidone and olanzapine will show greater benefits than conventional medications on assessments of social cognition, particularly affect perception and social perception.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosed with schizophrenia disorder by a DSM IV.
* Competent to sign informed consent
* No history of poor response to Risperdal and Zyprexa
* No organic brain disease

Exclusion Criteria:

* Mental retardation or any chronic medical illness which results in the patient not being appropriate for a switch to Risperdal or Zyprexa.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Dates: Start 2003-10; Study Completion 2006-03

CONTACTS AND LOCATIONS:
Locations (1):
- VA Greater Los Angeles Healthcare System, Los Angeles, California, United States

REFERENCES:
- [Derived] Sergi M, Green M, Widmark C, Reist C, Erhart S, Braff D, Kee K, Marder S, Mintz J. Social Cognition and Neurocognition: Effects of Risperidone, Olanzapine, and Haloperidol. Am J Psychiatry. 2007 Oct 1;164(10):1585-1592. doi: 10.1176/appi.ajp.2007.06091515. PMID 22688151
- [Derived] Sergi MJ, Green MF, Widmark C, Reist C, Erhart S, Braff DL, Kee KS, Marder SR, Mintz J. Social cognition [corrected] and neurocognition: effects of risperidone, olanzapine, and haloperidol. Am J Psychiatry. 2007 Oct;164(10):1585-92. doi: 10.1176/appi.ajp.2007.06091515. PMID 17898351